CLINICAL TRIAL: NCT02515968
Title: Comparison of Desflurane and Propofol on Quality of Recovery in Patients Undergoing Robotic or Laparoscopic Gastrectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The paper is about to publish on the same subject abroad, so the investigator decieded to stopped the study.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2015-0509
Record Dates: First submitted 2015-08-03; First posted 2015-08-05 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: General Anesthesia
MeSH Terms: interventions — Desflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Desflurane (Active Comparator): Anesthesia is maintained with desflurane during surgery.
  Interventions: Drug: Desflurane
- Propofol (Experimental): Anesthesia is maintained with propofol during surgery.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Desflurane — Anesthesia is maintained with desflurane in Desflurane group according to the randomly allocated groups.
  Arms: Desflurane
Drug: Propofol
  Other Names: Anesthesia is maintained with propofol in Propofol group according to the randomly allocated groups.
  Arms: Propofol

SUMMARY:
The purpose of this study is to investigate whether propofol can improve quality of recovery compared to desflurane in patients undergoing robotic or laparoscopic gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* adult patients aged over 20 yrs who are scheduled for laparoscopic or robotic gastrectomy, ASA 1 or 2.

Exclusion Criteria:

* patients with allergy to anesthetic agents
* body mass index more than 35 kg/m2
* pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Quality of recovery | Within 24 hours after the end of surgery
  The quality of recovery will be assessed with QoR-40 score.